CLINICAL TRIAL: NCT01238744
Title: Effect of Flaxseed Mucilage Drinks and Tablets on Satiety and Energy Intake
Brief Title: Flaxseed Mucilage and Satiety
Acronym: MUCISAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Copenhagen (Other)
Responsible Party: Mette Kristensen, Ass Prof, Department of Human Nutrition, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: B271
Record Dates: First submitted 2010-11-10; First posted 2010-11-11 (Estimated); Last update posted 2010-11-11 (Estimated); Status verified 2010-08

CONDITIONS: Appetite
MeSH Terms: interventions — Linseed Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Study I: control drink (Placebo Comparator)
  Interventions: Dietary Supplement: Control drink
- Study I: flaxseed drink (Experimental)
  Interventions: Dietary Supplement: Flaxseed drink
- Study II: flaxseed drink (Active Comparator)
  Interventions: Dietary Supplement: Flaxseed drink
- Study II: flaxseed tablets (Experimental)
  Interventions: Dietary Supplement: Flaxseed tablet

INTERVENTIONS:
Dietary Supplement: Flaxseed drink — Drink containing flaxseed mucilage
  Arms: Study I: flaxseed drink
Dietary Supplement: Flaxseed drink — Drink containing flaxseed mucilage
  Arms: Study II: flaxseed drink
Dietary Supplement: Flaxseed tablet — Tablets containing flaxseed mucilage consumed with a control drink
  Arms: Study II: flaxseed tablets
Dietary Supplement: Control drink — Control drink
  Arms: Study I: control drink

SUMMARY:
The effect of a single dose of flaxseed mucilage incorporated into either drinks or tablets will be tested in term of their effect on appetite sensation measured using visual analogue scales over 120 minutes and ad libitum energy intake hereafter in two studies.

DETAILED DESCRIPTION:
Study I:

Control drink vs. Flaxseed drink consumed and appetite sensation registered over 120 minutes. Hereafter energy intake was measured.

Study II:

Flaxseed drink vs. Flaxseed tablets+control drink consumed and appetite sensation registered over 120 minutes. Hereafter energy intake was measured.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults
* 18-40 years
* BMI 19-28

Exclusion Criteria:

* smoking
* pregnancy or lactation
* excessive exercise
* medication (oral contraceptives the only exception)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2009-08; Primary Completion 2010-08 (Actual); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Appetite sensation | 120 minutes
  Appetite sensation measured by visual analogue scales

SECONDARY OUTCOMES:
Energy intake | 120 minutes
  Ad libitum energy intake at the next meal